CLINICAL TRIAL: NCT01015664
Title: A Phase I/II Trial of the Combination of Cisplatin, Cetuximab, and Temsirolimus in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Combination of Cisplatin, Cetuximab and Temsirolimus in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Tennessee Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Jeffrey Allen, MD, University of Tennessee Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN0209
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — temsirolimus; Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: temsirolimus — 10, 15, or 25 mg IV over 30 minutes on Days 1, 8, 15 and 22
  Other Names: Torisel
Drug: cisplatin — 75 mg/m2 IV over 60 minutes on day 1
  Other Names: Platinol
Drug: cetuximab — 400 mg m2 on Day 1 of Cycle 1, then 250 mg/m2 IV over 60 minutes on Days 1, 8, 15, and 22
  Other Names: Erbitux

SUMMARY:
This study will accrue in two "phases". During the first "phase" of the study, the optimal dose of temsirolimus in combination with cisplatin and cetuximab will be determined. It is expected that between 9-12 patients will be needed for this dose finding phase. Once the optimal dose has been determined, an additional 41 patients will be enrolled in the second "phase" of the study. The primary purpose of second phase of the study is to learn what effects, good and/or bad, temsirolimus in combination with cisplatin and cetuximab has on recurrent or metastatic head and neck cancer.

Collection of additional blood and tissue specimens will make it possible to do special tests, which will provide us information about how tumors respond to the chemotherapy, how your body breaks down and processes the drug, how differences in the genetic makeup of each person affects how the drug may work and is processed in the body, and how the drug affects proteins and cells in the body. We hope to determine if results of the specialized tests done on blood will help to predict which patients are more likely to benefit from the use of the drugs used in this study.

DETAILED DESCRIPTION:
The epidermal growth factor receptor (EGFR) pathway is a key molecular pathway in the pathogenesis of SCCHN. Cetuximab, a therapy targeting the EGFR pathway, has shown great promise in SCCHN. The EXTREME study found that by combining cetuximab to a regimen of cisplatin and 5-fluorouracil, PFS could be extended to 5.6 months from 3.3 months, and that overall survival increased to 10.1 months versus 7.4 months. While this study proved a survival benefit with the addition of cetuximab, there were high rates of Grade 3 or 4 toxicities to the chemotherapy backbone of high dose cisplatin with 5-fluorouracil.

The mammalian target of rapamycin (mTOR) pathway is activated when conditions favor cellular growth and proliferation. The PI3K-Akt pathway is one of the key modulators in the activation of mTOR. Phosphorylated Akt is detected in the majority of SCCHN tumors by immunohistochemistry.

Temsirolimus is an mTOR inhibitor that has been shown to have a synergistic effect with cisplatin and carboplatin in other tumor models. Due to the minimal toxicities associated with temsirolimus in clinical studies to date, this is an ideal agent to use in combination with other chemotherapies.

There is limited experience for the combination of EGFR inhibitors and mTOR inhibitors in human subjects. These agents have been combined with a suggested synergistic effect in preclinical models of colon cancer xenografts and cell lines from non-small cell lung, pancreas, colon, and breast cancers. Cetuximab has been safely combined with everolimus (on oral mTOR inhibitor) in human subjects.

There is sufficient evidence to suggest that the addition of the mTOR inhibitor, temsirolimus, may increase both the cytotoxicity seen from platinum-based chemotherapy as well as augment the effect of EGFR pathway inhibition from cetuximab, and possibly provide clinical benefit of its own. It is hypothesized that the combination of cisplatin, cetuximab, and temsirolimus will be an effective, well tolerated regimen for patients with R/M SCCHN.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years of age and have a histologically confirmed diagnosis of R/M SCCHN which is no longer amenable to curative surgical or radiation therapy.
2. Patients must sign a written informed consent form and HIPAA statement.
3. Patients must undergo biopsy for confirmation of R/M disease within 6 weeks (42 days) of study entry and be willing and able to comply with peripheral blood collections for the purpose of correlative studies. Biopsy of primary or metastatic site(s) is allowed, provided the site has not been previously irradiated.
4. Patients must have measurable disease as defined by RECIST.
5. Patients must have ECOG PS 0 or 1.
6. Patients must have adequate hematologic function as defined by an ANC ≥ 1,500, hemoglobin ≥ 10 g/dL, and a platelet count ≥ 75,000 obtained within 14 days prior to treatment.
7. Patients must have adequate hepatic function as defined by a total bilirubin ≤ 1.5 mg/dL and AST (SGOT) and ALT (SGPT) ≤ 2 times the ULN obtained within 14 days prior to treatment.
8. Patients must have adequate renal function defined as a serum creatinine ≤ 1.5 mg/dL or calculated CrCl ≥ 55 mL/minute (calculations should be conducted using the Cockroft-Gault equation).
9. Patients must have adequate lipid control defined as a serum cholesterol ≤ 350 mg/dL and serum triglycerides ≤ 300 mg/dL obtained within 14 days prior to treatment.
10. Patients must not have received previous chemotherapy for the treatment of R/M SCCHN. Previous curative-intent treatment with chemotherapy, radiation therapy, chemoradiotherapy, or surgery for locoregional disease is allowed provided at least 3 months have elapsed since the completion of previous therapies and the patient has recovered from all treatment related toxicities.
11. Patients may have received prior radiation therapy for symptomatic sites of disease progression provided that ≥ 21 days have elapsed since treatment and the patient has recovered from any treatment related toxicities.
12. Males and females of reproductive potential must agree to use effective contraception for the duration of study participation.

Exclusion Criteria:

1. Patients with active or prior CNS metastases.
2. Patients with a history of previous hypersensitivity reaction to study drugs.
3. Patients with other active malignancies are excluded. Patients with a history of non-melanoma skin cancers, in-situ cervical cancer, definitively treated stage I or II cancers from which the patient is in remission, or a history of other malignancies from which the patient has been disease free for ≥ 5 years are permitted.
4. Concurrent therapy with any other anti-cancer treatments.
5. Ongoing or active clinically serious infection requiring IV antibiotics or active HIV infection.
6. Patients with a history of symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any medical condition that could compromise the safety of the patient.
7. Patients with, in the best judgment of the investigator, psychosocial, family, sociological, or geographical limitations which could impact the patient's ability to comply with study procedures.
8. Pregnant or lactating females.
9. Employees of the investigator or study center with direct involvement in this or other studies under the direction of the investigative team.
10. Patients currently taking any of the following medications are ineligible: phenytoin, carbamazepine, phenobarbitor, and/or rifampin as these are all strong Cyp3A4/5 inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Phase one - the outcome measure for determining the optimal dose will be determined by whether the subjects experience a dose limiting toxicity (DLT)
Phase 2 - the outcome measure of Progression-Free Survival is defined as the time from first treatment to the documented progression of disease or death, whichever comes first.

SECONDARY OUTCOMES:
Overall response rate is defined as the proportion of patients achieving any response (CR + PR) compared to the total patient population.
Disease control rate is defined as the proportion of patients who achieve a CR, PR, or SD (for ≥ 12 weeks) during study treatment compared to the total patient population.
Overall survival is defined as the time from first treatment to the time of death, regardless of cause.

CONTACTS AND LOCATIONS:
Overall Officials: Furhan Yunus, MD, Principal Investigator — University of Tennessee Cancer Institute
Locations (1):
- Boston Baskin Caner Foundation, Memphis, Tennessee, United States